CLINICAL TRIAL: NCT03896009
Title: MOMENTUM: A Randomized, Double-blind, Single-dose, Placebo-controlled Study to Assess the Efficacy and Safety of AXS-07 (Meloxicam and Rizatriptan) for the Acute Treatment of Migraine in Adults
Brief Title: Maximizing Outcomes in Treating Acute Migraine
Acronym: MOMENTUM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Axsome Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AXS-07-301
Record Dates: First submitted 2019-03-15; First posted 2019-03-29 (Actual); Results first posted 2023-08-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Migraine
Keywords: Migraine; AXS-07; Meloxicam; Rizatriptan; Axsome; Axsome Therapeutics; MoSEIC meloxicam
MeSH Terms: conditions — Migraine Disorders | interventions — rizatriptan; Meloxicam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- AXS-07 (Experimental): Taken once upon a qualifying migraine
  Interventions: Drug: AXS-07 (MoSEIC meloxicam and rizatriptan)
- Meloxicam (Active Comparator): Taken once upon a qualifying migraine
  Interventions: Drug: Meloxicam
- Rizatriptan (Active Comparator): Taken once upon a qualifying migraine
  Interventions: Drug: Rizatriptan
- Placebo (Placebo Comparator): Taken once upon a qualifying migraine
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AXS-07 (MoSEIC meloxicam and rizatriptan) — AXS-07 taken once upon onset of a qualifying migraine.
  Arms: AXS-07
Drug: Meloxicam — Meloxicam taken once upon onset of a qualifying migraine.
  Arms: Meloxicam
Drug: Rizatriptan — Rizatriptan taken once upon onset of a qualifying migraine.
  Arms: Rizatriptan
Drug: Placebo — Placebo taken once upon onset of a qualifying migraine.
  Arms: Placebo

SUMMARY:
AXS-07 is an oral, investigational medicine consisting of MoSEIC meloxicam and rizatriptan, which is being developed for the acute treatment of migraine with or without aura in adults. AXS-07 tablets are formulated to provide an enhanced rate of absorption of meloxicam. This study is designed to evaluate the efficacy and safety of AXS-07 compared to meloxicam, rizatriptan, and placebo for the treatment of a migraine attack.

This is a randomized, double-blind, 4-arm, parallel group, single-dose, placebo-controlled trial. Subjects who successfully complete screening and continue to meet all entry criteria will be randomly assigned to take one dose of either AXS-07, meloxicam, rizatriptan, or placebo upon the occurrence of a qualifying migraine.

ELIGIBILITY:
Key Inclusion Criteria:

* Has an established diagnosis of migraine with or without aura.
* Has experienced an inadequate response to prior acute treatments.

Key Exclusion Criteria:

* Has previously received any investigational drug or device or investigational therapy within 30 days before Screening.
* Pregnant, breastfeeding, or planning to become pregnant or breastfeed during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1594 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2019-12-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (83):
- United States (83):
  - Clinical Research Site, Birmingham, Alabama
  - Clinical Research Site, Mobile, Alabama
  - Clinical Research Site, Phoenix, Arizona
  - Clinical Research Site, Tempe, Arizona
  - Clinical Research Site, Little Rock, Arkansas
  - Clinical Research Site, Canoga Park, California
  - Clinical Research Site, Colton, California
  - Clinical Research Site, Culver City, California
  - Clinical Research Site, Encino, California
  - Clinical Research Site, Los Alamitos, California
  - Clinical Research Site, Los Angeles, California
  - Clinical Research Site, Oceanside, California
  - Clinical Research Site, Pomona, California
  - Clinical Research Site, Redlands, California
  - Clinical Research Site, Riverside, California
  - Clinical Research Site, San Diego, California
  - Clinical Research Site, Santa Monica, California
  - Clinical Research Site, Spring Valley, California
  - Clinical Research Site, Walnut Creek, California
  - Clinical Research Site, Waterbury, Connecticut
  - Clinical Research Site, Clermont, Florida
  - Clinical Research Site, DeLand, Florida
  - Clinical Research Site, Fernandina Beach, Florida
  - Clinical Research Site, Hallandale, Florida
  - Clinical Research Site, Hialeah, Florida
  - Clinical Research Site, Hollywood, Florida
  - Clinical Research Site, Jacksonville, Florida
  - Clinical Research Site, Lake City, Florida
  - Clinical Research Site, Lake Worth, Florida
  - Clinical Research Site, Miami, Florida
  - Clinical Research Site, Ocoee, Florida
  - Clinical Research Site, Orange City, Florida
  - Clinical Research Site, Orlando, Florida
  - Clinical Research Site, Ormond Beach, Florida
  - Clinical Research Site, South Miami, Florida
  - Clinical Research Site, Sunrise, Florida
  - Clinical Research Site, Tampa, Florida
  - Clinical Research Site, Atlanta, Georgia
  - Clinical Research Site, Stockbridge, Georgia
  - Clinical Research Site, Meridian, Idaho
  - Clinical Research Site, Evanston, Illinois
  - Clinical Research Site, Lenexa, Kansas
  - Clinical Research Site, Lexington, Kentucky
  - Clinical Research Site, Louisville, Kentucky
  - Clinical Research Site, New Orleans, Louisiana
  - Clinical Research Site, Boston, Massachusetts
  - Clinical Research Site, North Dartmouth, Massachusetts
  - Clinical Research Site, Watertown, Massachusetts
  - Clinical Research Site, Ann Arbor, Michigan
  - Clinical Research Site, Minneapolis, Minnesota
  - Clinical Research Site, Kansas City, Missouri
  - Clinical Research Site, Springfield, Missouri
  - Clinical Research Site, Las Vegas, Nevada
  - Clinical Research Site, Berlin, New Jersey
  - Clinical Research Site, Toms River, New Jersey
  - Clinical Research Site, Albuquerque, New Mexico
  - Clinical Research Site, Endwell, New York
  - Clinical Research Site, Manlius, New York
  - Clinical Research Site, New York, New York
  - Clinical Research Site, Rochester, New York
  - Clinical Research Site, The Bronx, New York
  - Clinical Research Site, Williamsville, New York
  - Clinical Research Site, High Point, North Carolina
  - Clinical Research Site, Wilmington, North Carolina
  - Clinical Research Site, Cincinnati, Ohio
  - Clinical Research Site, Cleveland, Ohio
  - Clinical Research Site, Dublin, Ohio
  - Clinical Research Site, Oklahoma City, Oklahoma
  - Clinical Research Site, Portland, Oregon
  - Clinical Research Site, Salem, Oregon
  - Clinical Research Site, Philadelphia, Pennsylvania
  - Clinical Research Site, Charleston, South Carolina
  - Clinical Research Site, Mt. Pleasant, South Carolina
  - Clinical Research Site, Knoxville, Tennessee
  - Clinical Research Site, Memphis, Tennessee
  - Clinical Research Site, Nashville, Tennessee
  - Clinical Research Site, Austin, Texas
  - Clinical Research Site, San Antonio, Texas
  - Clinical Research Site, Salt Lake City, Utah
  - Clinical Research Site, Charlottesville, Virginia
  - Clinical Research Site, Norfolk, Virginia
  - Clinical Research Site, Bellevue, Washington
  - Clinical Research Site, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Axsome Therapeutics Website — http://www.axsome.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AXS-07 | Meloxicam | Rizatriptan | Placebo
Started | 456 | 455 | 456 | 227
Completed | 441 | 433 | 434 | 218
Not Completed | 15 | 22 | 22 | 9

BASELINE CHARACTERISTICS:
Population: Safety Population includes all subjects who received study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | AXS-07 | Meloxicam | Rizatriptan | Placebo | Total
Number analyzed (Participants) | 441 | 433 | 434 | 218 | 1526
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.1 (11.64) | 41.0 (12.13) | 41.5 (10.75) | 41.0 (11.71) | 41.1 (11.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 357 | 363 | 366 | 185 | 1271
  Male | 84 | 70 | 68 | 33 | 255
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 1 | 2 | 0 | 7
  Asian | 9 | 10 | 6 | 4 | 29
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 76 | 88 | 84 | 48 | 296
  White | 345 | 330 | 332 | 160 | 1167
  More than one race | 3 | 4 | 5 | 4 | 16
  Unknown or Not Reported | 4 | 0 | 5 | 2 | 11

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Reporting Headache Pain Freedom
Description: Absence of headache pain. AXS-07 vs Placebo.
Time Frame: Hour 2 following dose administration
Population: ITT population consists of all randomized subjects who received study drug and had a qualifying migraine.
Measure: Count of Participants; unit: Participants
Arm/Group | AXS-07 | Placebo
Number analyzed (Participants) | 428 | 209
Participants | 85 | 14
Statistical Analysis 1: Comparison: AXS-07 vs Placebo; Test type: Superiority; p < 0.001, Chi-squared

2. Primary Outcome: Percentage of Subjects With Absence of Most Bothersome Symptom
Description: Absence of most bothersome symptom, defined at the onset of migraine. AXS-07 vs Placebo.
Time Frame: Hour 2 following dose administration
Population: ITT population consists of all randomized subjects who received study drug and had a qualifying migraine.
Measure: Count of Participants; unit: Participants
Arm/Group | AXS-07 | Placebo
Number analyzed (Participants) | 428 | 209
Participants | 158 | 51
Statistical Analysis 1: Comparison: AXS-07 vs Placebo; Test type: Superiority; p = 0.002, Chi-squared

ADVERSE EVENTS:
Time Frame: Adverse events were collected after administration of study drug through the final visit (up to 1 week). Any AE was monitored up to a maximum of 30 days after the final visit.
Description: Safety Population includes all subjects who received study drug.
Arm/Group | AXS-07 | Meloxicam | Rizatriptan | Placebo
All-Cause Mortality (participants affected / at risk) | 0/441 | 0/433 | 0/434 | 0/218
Serious Adverse Events (participants affected / at risk) | 1/441 | 0/433 | 0/434 | 0/218
Other Adverse Events (participants affected / at risk) | 49/441 | 50/433 | 67/434 | 13/218
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AXS-07 (N=441) | Meloxicam (N=433) | Rizatriptan (N=434) | Placebo (N=218)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AXS-07 (N=441) | Meloxicam (N=433) | Rizatriptan (N=434) | Placebo (N=218)
Nausea (Gastrointestinal disorders) | 12 (12) | 14 (15) | 21 (21) | 8 (8)
Dizziness (Nervous system disorders) | 7 (7) | 5 (5) | 9 (9) | 2 (2)
Somnolence (Nervous system disorders) | 6 (6) | 10 (10) | 9 (9) | 1 (1)
All Others, occurring in <1% of Subjects (General disorders) | 28 | 22 | 32 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-16): https://cdn.clinicaltrials.gov/large-docs/09/NCT03896009/Prot_SAP_000.pdf